CLINICAL TRIAL: NCT07279714
Title: Fisetin Intervention Study in Mild Alzheimer's Disease
Brief Title: Fisetin in Mild Alzheimer's Disease
Acronym: FIS-AD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6705
Record Dates: First submitted 2025-11-17; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer s Disease; Alzheimer Dementia; Alzheimer Dementia (AD); Alzheimer Disease; Mild Cognitive Disorder; Neurocognitive Disorders, Mild; Neurocognitive Disorder
Keywords: fisetin; alzheimer's disease; safety; tolerability
MeSH Terms: conditions — Alzheimer Disease; Neurocognitive Disorders | interventions — fisetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fisetin (Experimental)
  Interventions: Other: Fisetin

INTERVENTIONS:
Other: Fisetin — Fisetin 20mg/kg/day

SUMMARY:
This pilot study will evaluate the safety and tolerability of the natural health product, fisetin, in older adults with mild cognitive impairment or mild Alzheimer's disease dementia.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment due to Alzheimer's disease OR mild Alzheimer Dementia
* Moca score of 11 or higher
* Stable psychotropics and cognitive enhancing medications

Exclusion Criteria:

* Known hypersensitivity or allergy to fisetin
* Presence of any medical condition, or abnormal routine blood test, that the investigator believes would put the subject at risk or would preclude the patient from completing all aspects of the trial
* Unstable medical disorders
* Ongoing treatment for active infection with antibiotics/antifungals
* Ongoing treatment for cancer
* Active alcohol or substance use disorder
* Recent active bleeding
* Patients taking oral anticoagulants, anti-cancer, anti-seizure medications, or other medications that could have a significant interaction with fisetin
* Use within the last month of other senolytic supplements, antioxidant supplements, natural health products
* Other neurologic or neurodegenerative conditions impacting cognition
* Active Major Depressive Episode, active suicidal thoughts or psychosis
* Any thing that would preclude the ability to undergo an MRI scan

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability of fisetin) | 30 days
  Measured using AE reports

CONTACTS AND LOCATIONS:
Overall Officials: Krista Lanctôt, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided